CLINICAL TRIAL: NCT05923450
Title: Presence of Tumor Deposits is a Strong Indicator of Poor Outcome in Stage III Colorectal Cancers Undergoing Radical Surgery: Need for an Urgent Revision of the Staging System
Brief Title: Tumor Deposits in Colorectal Cancers
Acronym: TD
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Gennaro Galizia, Full Professor of Surgery, University of Campania Luigi Vanvitelli
Other Study IDs: Vanvitelli Naples
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Extranodal Extension
Keywords: tumor deposits; colorectal cancers; TNM staging system; ROC Curve
MeSH Terms: conditions — Extranodal Extension; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tumor Deposits: Colorectal cancers with and without tumor deposits, undergoing curative surgery and adjuvant chemotherapy
  Interventions: Procedure: Colorectal Resection

INTERVENTIONS:
Procedure: Colorectal Resection — Radical resection of colorectal cancer

SUMMARY:
Tumor deposits (TDs) are emerging as an adverse prognostic factor in colorectal cancers (CRCs), but they are quite ignored in the current staging system. Previous proposals to incorporate TDs in node stage or consider them distant metastases raised some doubt. The Authors propose a new staging system to optimize treatments.

DETAILED DESCRIPTION:
Tumor deposits (TDs) are emerging as an adverse prognostic factor in colorectal cancers (CRCs).In the current staging system TDs are somewhat neglected.

It has been proposed to add TD count to the number of metastatic lymph nodes or to consider TDs as distant metastases, but the scientific basis of these proposals seems dubious and not supported by robust statistical analyses.

The investigators supposed that splitting the three sub-stages of the stage III CRC according to absence or presence of TDs could be an easy and useful method to avoid the loss of crucial information. The proposed study will include 243 stage III CRC patients undergoing radical surgery and adjuvant chemotherapy. Each new substage, according to absence or presence of tumor deposits, will be analyzed with sophisticated statistical analysis (particularly the area-under-curve (AUC), calculated by the time-dependent receiver-operating-characteristic (ROC) curve for censored survival data) to individuate if this new staging does better the current one.

ELIGIBILITY:
Inclusion Criteria:

* colorectal cancers in stage III TNM undergoing radical surgery and adjuvant chemotherapy

Exclusion Criteria:

* Lynch syndrome
* Rectal Cancer undergoing neoadjuvant (radio)chemotherapy
* colorectal cancers without metastatic nodes
* metastatic colorectal cancers
* eligible patients refusing adjuvant chemotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: colorectal cancer patients with metastatic nodes undergoing radical surgery and adjuvant chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 243 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 5 years
  1 to 5 years overall survival
Disease-free Survival | 5 years
  1 to 5 years disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Gennaro Galizia, MD, Principal Investigator — University of Campania 'Luigi Vanvitelli'

IPD SHARING:
Plan to Share IPD: Yes
all data will be shared after publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: one month after publication
Access Criteria: email to gennaro.galizia@unicampania.it

REFERENCES:
- [Background] Galizia G, Lieto E, Auricchio A, Cardella F, Mabilia A, Podzemny V, Castellano P, Orditura M, Napolitano V. Naples Prognostic Score, Based on Nutritional and Inflammatory Status, is an Independent Predictor of Long-term Outcome in Patients Undergoing Surgery for Colorectal Cancer. Dis Colon Rectum. 2017 Dec;60(12):1273-1284. doi: 10.1097/DCR.0000000000000961. PMID 29112563
- [Result] Cervantes A, Adam R, Rosello S, Arnold D, Normanno N, Taieb J, Seligmann J, De Baere T, Osterlund P, Yoshino T, Martinelli E; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Metastatic colorectal cancer: ESMO Clinical Practice Guideline for diagnosis, treatment and follow-up. Ann Oncol. 2023 Jan;34(1):10-32. doi: 10.1016/j.annonc.2022.10.003. Epub 2022 Oct 25. No abstract available. PMID 36307056
- [Result] Pyo DH, Kim SH, Ha SY, Yun SH, Cho YB, Huh JW, Park YA, Shin JK, Lee WY, Kim HC. Revised Nodal Staging Integrating Tumor Deposit Counts With Positive Lymph Nodes in Patients With Stage III Colon Cancer. Ann Surg. 2023 Apr 1;277(4):e825-e831. doi: 10.1097/SLA.0000000000005355. Epub 2021 Dec 23. PMID 34954753
- [Result] Khan H, Radomski SN, Siddiqi A, Zhou N, Paneitz DC, Johnston FM, Greer JB. Tumor deposits are associated with a higher risk of peritoneal disease in non-metastatic colorectal cancer patients. J Surg Oncol. 2023 May;127(6):975-982. doi: 10.1002/jso.27207. Epub 2023 Feb 15. PMID 36790093
- [Derived] Lieto E, Auricchio A, Ronchi A, Del Sorbo G, Panarese I, Ferraraccio F, De Vita F, Galizia G, Cardella F. Presence of tumor deposits is a strong indicator of poor outcome in patients with stage III colorectal cancers undergoing radical surgery. J Gastrointest Surg. 2024 Jan;28(1):47-56. doi: 10.1016/j.gassur.2023.11.003. PMID 38353074